CLINICAL TRIAL: NCT04634656
Title: Neuroprotective Effects of Lidocaine on Early Postoperative Cognitive Dysfunction in Patients Undergoing Shoulder Arthroscopy With Beach Chair Position: a Randomized Trial
Brief Title: Lidocaine on Early Cognitive Dysfunction in Shoulder Arthroscopy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM 2020
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Cognitive Dysfunction, Postoperative
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Active Comparator): Patients will receive lidocaine in a loading dose of 1 mg/ kg diluted in 10 ml of normal saline that will be infused over 5 minutes after induction of anesthesia then followed by a continuous infusion at 1.5 mg/ kg/ h diluted in normal saline to a volume of 50 ml until the end of surgery.
  Interventions: Drug: Lidocaine
- Group C (Placebo Comparator): Patients will receive normal saline after induction of anesthesia with the same volume and rate changes as lidocaine group until the end of surgery.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Patients will receive lidocaine in a loading dose of 1 mg/ kg diluted in 10 ml of normal saline that will be infused over 5 minutes after induction of anesthesia then followed by a continuous infusion at 1.5 mg/ kg/ h diluted in normal saline to a volume of 50 ml until the end of surgery
  Other Names: Xylocaine
  Arms: Group L
Drug: Normal saline — Patients will receive normal saline after induction of anesthesia with the same volume and rate changes as lidocaine group until the end of surgery
  Arms: Group C

SUMMARY:
The beach chair position (BCP) combined with deliberate hypotension impair cerebral perfusion pressure and oxygenation during arthroscopic shoulder surgeries and produce cerebral ischemia.

DETAILED DESCRIPTION:
Arthroscopic diagnosis and treatment of shoulder disorders have replaced open procedure as the primary treatment method. The beach chair (BCP) and lateral decubitus (LDP) positions are both considered as reliable techniques for performing effective arthroscopic shoulder surgeries. The usage of BCP for shoulder arthroscopic operations started from early 1980s.

The advantages of BCP include lack of brachial plexus strain, good intra-articular visualization, with the ease of conversion to an open approach if required.

The BCP combined with deliberate hypotension has been used to decrease intraoperative blood loss and allow a relatively blood-free surgical field. However, this combination has the risk to impair cerebral perfusion pressure and oxygenation during surgery and produce cerebral ischemia.

Lidocaine, a commonly used local anesthetic and class IB antiarrhythmic drug, that readily crosses the blood - brain barrier. Evans et al. initially reported cerebral protection of lidocaine in a feline model of cerebral arterial gas embolism. Later on, the effects of lidocaine on perioperative neuroprotection were detected. However, the mechanisms underlying lidocaine treatment-induced neuroprotection remain incompletely understood.

Lidocaine may provide cerebral protection through many mechanisms, including decreasing the cerebral metabolic rate, decelerating the ischemic transmembrane ion shift, and reducing the ischemic excitotoxin release.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective arthroscopic shoulder surgery under general anesthesia in beach chair position (BCP),
* Age 20 to 65 years old.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score < 23 before surgery
* History of neurological disease (such as previous episodes of cerebral ischemia or stroke).
* History of psychological disorder
* Suspected history of adverse reactions to lidocaine
* Drug or alcohol abuse
* History of diabetes mellitus, sever hypertension, severe anemia, hepatic or renal dysfunction
* Unwillingness to comply with protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-11-10 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative cognitive function | 3 days after surgery
  Assessed using Mini-Mental State Examination (MMSE) test

CONTACTS AND LOCATIONS:
Overall Officials: Seham M Moeen, MD, Principal Investigator — Assiut University
Locations (1):
- Seham Mohamed Moeen, Asyut, Asyut Governorate, Egypt